CLINICAL TRIAL: NCT04104893
Title: A Phase 2 Study of a Checkpoint Inhibitor in Men With Progressive Metastatic Castrate Resistant Prostate Cancer Characterized by a Mismatch Repair Deficiency or Biallelic CDK12 Inactivation
Brief Title: A Study of CHeckpoint Inhibitors in Men With prOgressive Metastatic Castrate Resistant Prostate Cancer Characterized by a Mismatch Repair Deficiency or Biallelic CDK12 Inactivation
Acronym: CHOMP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSDR-003-18F; CX002006 (Other Grant/Funding Number: CSR&D)
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Metastatic Prostate Cancer; Pembrolizumab; Checkpoint Inhibitor; Mismatch Repair Deficiency; CDK12
MeSH Terms: conditions — Prostatic Neoplasms; Turcot syndrome | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients with either a mismatch repair deficiency or biallelic inactivation of CDK12 in their tumor are eligible for this study. Patients with these mutations will be identified primarily through standard of care genetic testing with either archival tissue or blood. Once enrolled the patient will undergo a biopsy of a metastatic lesion (baseline biopsy) to identify molecular correlates.
  Pembrolizumab will be administered at a starting dose of 200 mg intravenously every 3 weeks until disease progression or unacceptable toxicity. During the treatment, patients will either simultaneously receive a GnRH analogue or undergo a bilateral orchiectomy prior to treatment to maintain a castrate level of testosterone ( 50 ng/dl). At progression, patients will undergo a second biopsy of the same metastatic lesion of the baseline biopsy. The baseline (pre-treatment) and at-progression biopsies will be used for correlative analyses to determine the efficacy of pembrolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): This is a single-arm, open-label study of the checkpoint inhibitor, pembrolizumab, in Veterans with mCRPC who have progressed on at least 1 prior novel androgen receptor (AR) signaling inhibitor, inclusive of abiraterone acetate, enzalutamide, apalutamide, and darolutamide. In addition to progressive mCRPC, a patient must have a somatic tumor mutation characterized by dMMR or CDK12-/- detected by next generation sequencing (NGS). Patients enrolled in this study will be treated with pembrolizumab at the FDA approved dosage of 200 mg intravenously every 3 weeks (21 days) until disease progression or unacceptable toxicity. During study, patients will maintain a castrate level of testosterone, = 50 ng/dL by ongoing treatment with a GnRH analogue or prior bilateral orchiectomy. Prior to initiating treatment with pembrolizumab, patients will undergo a baseline biopsy of a metastatic lesion. An additional biopsy of a metastatic lesion at the time of progression will be encouraged as well.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a programmed death receptor-1 (PD 1)-blocking antibody. Pembrolizumab is a humanized monoclonal IgG4 kappa antibody with an approximate molecular weight of 149 kDa. Pembrolizumab is produced in recombinant Chinese hamster ovary (CHO) cells.
  Other Names: Keytruda

SUMMARY:
The primary objective is to assess the activity and efficacy of pembrolizumab, a checkpoint inhibitor, in Veterans with metastatic castration-resistant prostate cancer (mCRPC) characterized by either mismatch repair deficiency (dMMR) or biallelic inactivation of CDK12 (CDK12-/-). The secondary objectives involve determining the frequency with which dMMR and CDK12-/- occur in this patient population, as well as the effects of pembrolizumab on various clinical endpoints (time to PSA progression, maximal PSA response, time to initiation of alternative anti-neoplastic therapy, time to radiographic progression, overall survival, and safety and tolerability). Lastly, the study will compare the pre-treatment and at-progression metastatic tumor biopsies to investigate the molecular correlates of resistance and sensitivity to pembrolizumab via RNA-sequencing, exome-sequencing, selected protein analyses, and multiplexed immunofluorescence.

DETAILED DESCRIPTION:
Research Plan:

This is a single-arm, open-label phase II study that examines the response rate of pembrolizumab in metastatic castration-resistant prostate cancer (mCRPC) patients who have either a mismatch repair deficiency (dMMR) or a biallelic inactivation of CDK12 (CDK12-/-). The study will enroll mCRPC patients who have the selected genetic mutation and at least one metastatic lesion that is amendable to biopsy. All patients must have progressed on at least one prior line of mCRPC therapy, such as abiraterone acetate or enzalutamide. Eligible patients will undergo at least 12 weeks (4 cycles) of pembrolizumab (200 mg IV).

Methodology:

Patients with either a mismatch repair deficiency or biallelic inactivation of CDK12 in their tumor are eligible for this study. If the patient has progressed on at least one prior therapy for mCRPC, including abiraterone acetate or enzalutamide, he is eligible to begin genetic screening. Patients with these mutations will be identified primarily through standard of care genetic testing with either archival tissue or blood. Specimens will be sent to VA approved vendors for genetic testing to determine if the patient has the necessary mutations to receive the study drug (pembrolizumab). If eligible, the patient will sign the Main Treatment ICF and proceed with the screening procedures. Once enrolled the patient will undergo a biopsy of a metastatic lesion (baseline biopsy) to identify molecular correlates. If the patient does not have any archival tissue or blood to be used to identify genetic mutations, the biopsy of a metastatic lesion will be used to both identify genetic mutations and to identify molecular correlates.

When the patient has met all the eligibility criteria, he will receive pembrolizumab. Pembrolizumab will be administered at a starting dose of 200 mg intravenously every 3 weeks until disease progression or unacceptable toxicity. During the treatment, patients will either simultaneously receive a GnRH analogue or undergo a bilateral orchiectomy prior to treatment to maintain a castrate level of testosterone ( 50 ng/dl). At progression, patients will undergo a second biopsy of the same metastatic lesion of the baseline biopsy. The baseline (pre-treatment) and at-progression biopsies will be used for correlative analyses to determine the efficacy of pembrolizumab.

Note: after the testing process is complete, Oncoplex will return any remaining sample back to the Department of Pathology at the West LA VA Medical Center. These specimens will be stored in Dr. Matthew Rettig's biorepository on site for analysis and future research.

Results:

Since this is a new study, the results have not yet been obtained. The primary endpoint of this study is to measure the objective response rate, radiographic progression free survival at 6 months, and decline in PSA of 50% or more 12 weeks of therapy.

Clinical Significance:

There are 230,000 new incidences of prostate cancer and 30,000 deaths from prostate cancer per year in the US. It is the second most common cause of death in American men. Importantly, prostate cancer is diagnosed in more than 12,000 US Veterans each year, representing nearly one third of all cancer diagnoses in Veterans.

Metastatic prostate cancer is incurable, and its treatment is palliative. However, many Veterans with metastatic castration-resistant prostate cancer (mCRPC) progress despite experiencing some clinical benefit from hormonal therapy and chemotherapy. As a result, novel therapies that provide a robust clinical benefit and have a good safety profile are needed for these patients.

Immunotherapies, such as checkpoint inhibitor, for mCRPC patients that have either a mismatch repair deficiency (dMMR) or a biallelic inactivation of CDK12 (CDK12-/-) is an attractive therapy, especially since therapies involving checkpoint inhibitors have exhibited significant improvements in patients with advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and many other cancers. The results of this study will establish the ideal subset of mCRPC patients who will benefit from the study drug. Importantly, the correlative studies will provide critical insight into the mechanisms of primary and acquired resistance that occur despite selection of patients with CDK12-/- or dMMR. This result can inform further selection of patients for checkpoint inhibition, as well as identify other potential therapies that can be co-administered with pembrolizumab to prevent or overcome resistance to checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older at the time the Informed Consent is signed.
* The subject (or legally acceptable representative if applicable) must provide written informed consent for the trial.
* Pathologic diagnosis of prostate cancer of adenocarcinoma or small cell histology.
* Metastatic disease as documented by technetium-99m (99mTc) bone scan or metastatic lesions by computed tomography (CT) or magnetic resonance imaging (MRI) scans (visceral or lymph node disease). CT-portion of FDG-PET/CT or scan may be used for eligibility. NaF PET-CT is an alternative to 99mTc bone scan. If lymph node metastasis is the only evidence of metastatic disease, it must be 1.5 cm in short axis and above the level of the iliac bifurcation. Imaging studies for the purpose of determining eligibility must be completed within 60 days of Day 1.
* Progressive castration resistant prostate cancer as defined by serum testosterone < 50 ng/mL and one of the following:

  * PSA progression confirmed per Prostate Cancer Clinical Trials Working Group (PCWG3),
  * Radiographic progression of soft tissues according to Response Evaluation Criteria in Solid Tumors, version 1.1 (iRECIST 1.1) modified based on PCWG3, or radiographic progression of bone according to PCWG3.
* Prior use of a novel AR signaling inhibitor for 4 weeks, including abiraterone acetate plus prednisone/prednisolone, enzalutamide, apalutamide, and/or darolutamide.

NOTE: These AR signaling inhibitors may have been used for mCSPC, M0CRPC, and/or mCRPC.

* Ongoing surgical or medical castration, with testosterone levels of <50 ng/dL. If the subject is being treated with GnRH analogs (subject who has not undergone bilateral orchiectomy), this therapy must have been initiated at least 30 weeks prior to initiation of pembrolizumab and must be continued throughout the study.
* ECOG PS grade of 0-1.
* Metastatic lesion that is amenable to biopsy and performed within 180 days of Day 1.
* dMMR or CDK12-/- as determined by somatic tumor DNA NGS.

  * Either monoallelic or biallelic inactivation of CDK12 on NGS is considered sufficient for eligibility purposes.
  * MMR genes include: MLH1, MSH2, MLH3, PMS1, MSH6, and PMS2.
  * dMMR is established by MSI-H on NGS. However, for "weak" MMR genes, inclusive of PMS2 and MSH6, monoallelic inactivation will be allowed for eligibility purposes if and only if there is at least MSI-low or hypermutation that is concomitantly present.
  * If there is biallelic inactivation of "strong" MMR genes (MLH1 and MSH2), then patients must manifest MSI-H. However, if the tumor DNA utilized for MSI analysis was obtained > 6 months prior to NGS, then the NGS should be repeated to determine if MSI-H has developed. Monoallelic inactivation of "strong" MMR genes will be allowed if MSI-H is present; in this scenario, it is presumed that biallelic inactivation is present but the second inactivating event was not detected due to technical issues such as low sensitivity for copy loss.
* Adequate organ function:

  * Hemoglobin (hgb) > 9.0 g/dL,
  * Absolute neutrophil count (ANC) > 1500/ uL,
  * Platelets > 100,000/ uL,
  * Total bilirubin 1.5 x ULN OR direct bilirubin ULN for participants with total bilirubin levels >1.5 x ULN
  * ALT and AST 2.5 x ULN ( 5 x ULN for participants with liver metastases) (Child-Pugh class A and B allowed; Child-Pugh class C is excluded).
  * Creatinine < (2.0 mg/dL) during screening evaluation (>2.0 is allowed if EGFR >30 mL/min/1.73 m2).
* Subject must agree to use contraception during the treatment period plus an additional 120 days after the last dose of study treatment and must refrain from donating sperm during this period.

Exclusion Criteria:

* Brain metastases.
* Prior treatment with an anti-PD1, anti-PDL1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Anti-neoplastic therapies for prostate cancer must be completed > 2 weeks prior to Day 1 (initiation of pembrolizumab); chemotherapy must be completed > 4 weeks prior to Day 1.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to [randomization /allocation].

Note: Participants must have recovered from all AEs due to previous therapies to Grade 1 or baseline. Participants with Grade 2 neuropathy may be eligible.

* Herbal and non-herbal products that may decrease PSA levels other than medical castration and megestrol (up to 40 mg/day is allowed) for hot flashes.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation ( 2 weeks of radiotherapy) to non-CNS disease.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* If a subject has undergone major surgery, they must have recovered adequately from the toxicities or complications from the intervention within 4 weeks prior to starting therapy.
* History of non-prostate active malignancy requiring treatment in the 24 months prior to Day 1 except for non-muscle invasive urothelial cancer and non-melanoma skin cancer.
* Active infection or conditions requiring treatment with antibiotics.
* Immunosuppressive doses of systemic medications, such as corticosteroids (doses > 10 mg/day prednisone or equivalent), within 2 weeks of Day 1.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Active autoimmune disease or a documented history of autoimmune disease that requires immunosuppressive medications within the last two years (e.g., chronic steroids, methotrexate, tacrolimus, etc.).
* Active or chronic hepatitis B or hepatitis C disease as determined by hepatitis B surface antigen (HBsAg), hepatitis B core antibody, or hepatitis C antibody (anti-HCV) positivity at screening. If positive, further testing of quantitative levels to rule out active infection is required.
* History of positive test for human immunodeficiency virus (HIV). NOTE: Hepatitis B and C and HIV testing is NOT required during screening.
* Vaccinated with a live vaccine within 30 days of enrollment.
* Has severe hypersensitivity ( Grade 3) to pembrolizumab and/or any of its excipients.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subject is planning to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study involves the treatment of patients with metastatic castration resistant prostate cancer with Pembrolizumab. Since only men have prostates, our study will be limited to only enrolling male subjects.
Enrollment: 40 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PSA Decline | 12 weeks of therapy
  Decline in PSA of 50% or more (PSA50) 12 weeks of therapy (ng/mL)
Objective Response Rate | First day of Pembrolizumab administration to 6 months after
  Objective response in measurable disease by immunotherapy response criteria (iRECIST) or radiographic progression free survival (rPFS) after 6 months of therapy.

SECONDARY OUTCOMES:
Time to Progression of Disease | Date of enrollment to the date of the last patient in plus one year after
  * Time to PSA progression
  * Time to initiation of alternative anti-neoplastic therapy,
  * Time to radiographic progression
Overall Survival | From enrollment until death assessed up to 36 months
  The overall survival rate measured as time from enrollment until death.
Maximum PSA Response | Date of Enrollement to the date of the last patient in plus one year after
  Maximal PSA response (ng/mL)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Date of first patient in to the date of the last patient in plus one year after
  See what the safety and tolerability of Pembrolizumab on patients with prostate cancer is by assessing adverse and serious adverse events that each patient experiences.

OTHER OUTCOMES:
Identification of Molecular Correlates and Biomarkers of Resistance and Sensitivity to Pembrolizumab | Date of enrollment to the date of the last patient in plus one year after
  We will investigate and identify molecular correlates and biomarkers of resistance and sensitivity to pembrolizumab using baseline and at-progression metastatic tumor biopsies. Molecular correlates will be assessed by RNA-seq, exome-seq, selected protein analyses, and multiplexed immunofluorescence for immune cells. Whenever possible, we will attempt to validate tissue based biomarkers in peripheral blood specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B. Rettig, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (13):
- United States (13):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
None of the biospecimens will be destroyed. Unused specimens will be used for future research to access clinical data indefinitely. Subjects can request to have all of their specimens destroyed at the end of the study. The research blood and tumor tissue specimens will not be marked with any personal identifiers. As soon as they are collected by a study personnel, the samples will be labeled with a code. The key to the code will remain locked in the research office that is only accessed by study personnel. Only coded specimens will be sent to commercial vendors and VA GLAHS in West LA.
  The study investigators will perform research testing on their tissue specimens that is independent of the genetic analysis to be performed at commercial vendor. There are no plans to share the results of other testing performed on their specimens. These results are only for research purposes. However, certain exploratory biomarker test results may be shared with the subject.